CLINICAL TRIAL: NCT05535660
Title: Lipid Profiles as Predictor of Adverse Maternal and Neonatal Outcomes: A Pilot Study
Brief Title: Lipid Profile as Predictor of Adverse Maternal and Neonatal Outcomes: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Samsiya Ona, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-21-01936-MOD002
Record Dates: First submitted 2022-08-19; First posted 2022-09-10 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Hyperlipidemia; Pregnancy
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- LGA neonates: Researchers will compare lipid levels in large for gestational age (LGA) and non-LGA neonates.
  Interventions: Diagnostic Test: Lipid panel
- non-LGA neonates: Researchers will compare lipid levels in large for gestational age (LGA) and non-LGA neonates.
  Interventions: Diagnostic Test: Lipid panel

INTERVENTIONS:
Diagnostic Test: Lipid panel — fasting blood draw to examine concentrations of lipids in maternal blood during pregnancy

SUMMARY:
The purpose of this study is to ascertain lipid profiles during pregnancy, specifically during the 24-28 week gestation and again near term at 36 weeks gestation. The research team are investigating whether lipid profiles can predict adverse maternal and neonatal outcomes.

DETAILED DESCRIPTION:
The purpose of this research is to investigate whether lipids profiles during pregnancy impact LGA and other adverse outcomes in pregnancy. Participants will have blood drawn twice; the first blood work is a fasting blood draw (separate blood draw) on the same day but preceding the standard glucose test. The second blood draw is drawn at the time of routine clinical care (third trimester blood work).

Patients will be approached at the time of the anatomy ultrasound for participation. If they consent to participate they will have a FASTING lipid panel drawn at the time of their 24-28w GCT and again at the time of their 36w third trimester labs. Patients will receive a reminder call prior to scheduled 24-28 week appointment for fasting instructions.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Ages 18-45
* Presentation to prenatal care by the 2nd trimester
* Prenatal care at Mount Sinai Hospital
* Anticipated delivery at Mount Sinai Hospital

Exclusion Criteria:

* Multiple gestations
* Preexisting hyperlipidemia
* Preexisting diabetes
* Delayed presentation to prenatal care after the 2nd trimester 5. Prenatal care or delivery outside of Mount Sinai Health System

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant individuals without preexisting hyperlipidemia
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Neonatal birthweight | at birth, day 1
  Neonatal birthweight will be classified as large for gestational age (LGA) or non-LGA

SECONDARY OUTCOMES:
Number of participants with preeclampsia | at birth, day 1
Number of participants with gestational diabetes | at birth, day 1
Total Cholesterol | at 24-28 weeks gestation
  Total Cholesterol obtained while fasting at 24-28 weeks gestation. Different blood tests can be done to measure each type of cholesterol. Total cholesterol level measures all types of cholesterol in the blood.
Total Cholesterol | at 36 weeks gestation
  Total Cholesterol obtained while fasting at 36 weeks gestation. Different blood tests can be done to measure each type of cholesterol. Total cholesterol level measures all types of cholesterol in the blood.
High-Density Lipoprotein Cholesterol (HDL) | at 24-28 weeks gestation
  High-Density Lipoprotein Cholesterol (HDL) obtained while fasting at 24-28 weeks. HDL helps keep arteries open and reduces the risk for heart attack. High levels of HDL may be nearly as protective for the heart as low levels of LDL
High-Density Lipoprotein Cholesterol (HDL) | at 36 weeks gestation
  High-Density Lipoprotein Cholesterol (HDL) obtained while fasting at 36 weeks. HDL helps keep arteries open and reduces the risk for heart attack. High levels of HDL may be nearly as protective for the heart as low levels of LDL
Triglycerides | at 24-28 weeks gestation
  Triglycerides obtained while fasting at 24-28 weeks gestation. Triglycerides interact with HDL cholesterol in such a way that HDL levels fall as triglyceride levels rise. High triglyceride levels are also associated with the inflammatory response -- the harmful effect of an overactive immune system that can cause considerable damage to cells and tissues, including the arteries.
Triglycerides | at 36 weeks gestation
  Triglycerides obtained while fasting at 36 weeks gestation. Triglycerides interact with HDL cholesterol in such a way that HDL levels fall as triglyceride levels rise. High triglyceride levels are also associated with the inflammatory response -- the harmful effect of an overactive immune system that can cause considerable damage to cells and tissues, including the arteries.
Low-Density Lipoprotein Cholesterol (LDL) | at 24-26 weeks gestation
  Low-Density Lipoprotein Cholesterol (LDL) obtained while fasting at 24-28 weeks gestation. Low-density lipoprotein (LDL) transports about 75% of the blood's cholesterol to the body's cells. Heart disease is least likely to occur among people with the lowest LDL levels. Lowering LDL is the primary goal of cholesterol drug and lifestyle therapy.
Low-Density Lipoprotein Cholesterol (LDL) | at 36 weeks gestation
  Low-Density Lipoprotein Cholesterol (LDL) obtained while fasting at 36 weeks gestation. Low-density lipoprotein (LDL) transports about 75% of the blood's cholesterol to the body's cells. Heart disease is least likely to occur among people with the lowest LDL levels. Lowering LDL is the primary goal of cholesterol drug and lifestyle therapy.
Very-low-density Lipoprotein Cholesterol (VLDL) | at 24-26 weeks gestation
  Very-low-density Lipoprotein Cholesterol (VLDL) obtained while fasting at 24-28 weeks gestation. VLDL is one of the three main types of lipoproteins. Lipoproteins are made up of cholesterol, triglycerides, and proteins. They move cholesterol, triglycerides, and other lipids (fats) around the body.
Very-low-density Lipoprotein Cholesterol (VLDL) | at 36 weeks gestation
  Very-low-density Lipoprotein Cholesterol (VLDL) obtained while fasting at 36 weeks gestation. VLDL is one of the three main types of lipoproteins. Lipoproteins are made up of cholesterol, triglycerides, and proteins. They move cholesterol, triglycerides, and other lipids (fats) around the body.
Total Cholesterol/HDL Ratio | at 24-26 weeks gestation
  Total Cholesterol/HDL Ratio obtained while fasting at 24-28 weeks gestation. The total cholesterol /HDL ratio is the proportion of one type of cholesterol to all the other cholesterol in the blood. Total cholesterol includes three substances HDL, LDL, and VLDL. Higher ratios indicate greater risk of heart coronary heart disease.
Total Cholesterol/HDL Ratio | at 36 weeks gestation
  Total Cholesterol/HDL Ratio obtained while fasting at 36 weeks gestation. The total cholesterol /HDL ratio is the proportion of one type of cholesterol to all the other cholesterol in the blood. Total cholesterol includes three substances HDL, LDL, and VLDL. Higher ratios indicate greater risk of heart coronary heart disease.

CONTACTS AND LOCATIONS:
Overall Officials: Samsiya Ona, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai OBGYN Faculty Practice Associates, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study.

DOCUMENTS (1):
  • Informed Consent Form (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT05535660/ICF_000.pdf